CLINICAL TRIAL: NCT00305695
Title: A Phase II Randomized Study of the Effect of Zoledronic Acid Versus Observation on Bone Mineral Density of the Lumbar Spine in Women Who Elect to Undergo Surgery That Results in Removal of Both Ovaries
Brief Title: Zoledronate or Observation in Maintaining Bone Mineral Density in Patients Who Are Undergoing Surgery to Remove Both Ovaries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GOG-0215; NCI-2009-00589 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-P6966; NOVARTIS-GOG-0215; CDR0000462217; NCI-06-C-0204; GOG-0215 (Other: Gynecologic Oncology Group); GOG-0215 (Other: DCP); GOG-0215 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome; Osteoporosis; Ovarian Carcinoma
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Osteoporosis; Ovarian Neoplasms | interventions — Zoledronic Acid

ARMS (2):
- Arm I (zoledroic acid) (Experimental): Beginning 60-90 days after surgery, patients receive zoledronate IV over 15 minutes once in months 3, 9, and 15.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Zoledronic Acid
- Arm II (clinical observation) (No Intervention): Patients are observed for 18 months after surgery.

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm I (zoledroic acid)
Drug: Zoledronic Acid — Given IV
  Other Names: [1-Hydroxy-2-(1H-imidazol-1-yl)ethylidene]bisphosphonic Acid; CGP 42446; CGP42446A; NDC-Zoledronate; Reclast; ZOL 446; Zometa
  Arms: Arm I (zoledroic acid)

SUMMARY:
This randomized phase II trial is studying zoledronate to see how well it works compared to observation in maintaining bone mineral density in patients who are undergoing surgery to remove both ovaries. Zoledronate may prevent bone loss in patients who are undergoing surgery to remove the ovaries.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the effect of zoledronate vs observation on bone loss associated with surgery (at a minimum, any surgical procedure that results in removal of both ovaries) in patients undergoing excision of both ovaries.

SECONDARY OBJECTIVE:

I. Compare the change in bone mineral density of the bilateral hip in patients treated with these regimens.

TERTIARY OBJECTIVE:

I. Compare the effect of zoledronate vs observation on biochemical markers of bone resorption and bone formation (N-telopeptide and bone specific alkaline phosphatase) during 1 year of treatment.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

All patients undergo surgery, with removal of both ovaries, in month 1. All patients are requested to take calcium supplements twice daily and a multivitamin containing vitamin D once daily beginning in month 1 and continuing for up to 18 months.

ARM I: Beginning 60-90 days after surgery, patients receive zoledronate IV over 15 minutes once in months 3, 9, and 15.

ARM II: Patients are observed for 18 months after surgery.

In both arms, patients complete physical activity questionnaires at baseline and in months 3, 9, 15, and 18. Patients undergo bone mineral density test of lumbar spine and total hip at baseline and in months 9 and 18. Patients also undergo blood collection at baseline and periodically during the study for biomarker studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have elected to undergo, or who have undergone (within 8 weeks) a surgical procedure that results (at minimum) in the absence of both ovaries

  * Patients enrolled in the screening arm of GOG-0199 who decide to undergo surgery are potentially eligible for GOG-0215
* Baseline bone mass density (BMD) T-Score ? -1.5 (no more than 1.5 standard deviation below the mean value for young adults) on both the total lumbar spine (L1-L4 region, not individual bones) and bilateral hip
* Patients who had/have at least 1 intact ovary at the time of surgery are eligible
* No prior distant metastatic malignant disease within the past 5 years

  * Patients treated for stage M1 (any T, any N) diagnosis in the past 5 years are ineligible
  * Patients who achieved a complete response after treatment for rM0 (any T, any N) within the past 5 years are eligible
* Premenopausal*

  * Last menstrual cycle occurred < 12 months prior to study enrollment
* GOG performance status 0-2
* Creatinine clearance > 60 mL/min
* No clinical or radiological evidence of existing fracture of the lumbar spine or bilateral hip
* No history of hip of spine fracture with low-intensity trauma or not associated with trauma
* No uncontrolled seizure disorder associated with falls
* No diseases that influence bone metabolism, including any of the following:

  * Paget?s disease
  * Osteogenesis imperfecta
  * Uncontrolled thyroid or parathyroid dysfunction within 12 months prior to study entry
* No other nonmalignant systemic disease, including any of the following:

  * Uncontrolled infection
  * Uncontrolled type 2 diabetes mellitus
  * Cardiovascular, renal, hepatic, or lung disease that would prevent prolonged follow-up

    * History of thrombosis or thromboembolism allowed
* No known HIV positivity
* No known hypersensitivity to zoledronate or other bisphosphonates
* No psychiatric, psychological, or other conditions that prevent fully informed consent
* No other active malignancy except nonmelanoma skin cancer
* No history of any medical condition that places the patient at risk for donating blood for research purposes (e.g., chronic infectious diseases, sever anemia, or hemophilia)
* Not pregnant
* Negative pregnancy test
* No current active dental problems, including any of the following:

  * Infection of the teeth or jawbone (maxilla or mandible)
  * Dental or fixture trauma
  * Current or prior diagnosis of osteonecrosis of the jaw
  * Exposed bone in the mouth
  * Slow healing after dental procedures
* No recent (within 6 weeks) or planned dental or jaw surgery (e.g., extraction or implants)
* No prior treatment for osteoporosis
* No adjuvant radiotherapy within the past 31 days
* No chemotherapy within the past 30 days
* No prior surgery to the hip or spine
* No prior systemic sodium fluoride for > 3 months during the past 2 years
* No more than 30 days use in the past 12 months and no concurrent tamoxifen, raloxifene, or any other selective estrogen-receptor modulator (SERM)
* More than 12 months since prior and no concurrent endocrine therapy

  * Insulin and/or oral antidiabetic medications allowed
  * Thyroid hormone replacement allowed
* More than 12 months since prior and no concurrent estrogen or hormone replacement therapy (estrogen plus progesterone or estrogen alone)

  * Prior or concurrent oral contraceptives allowed
  * Systemic (oral) hormone replacement therapy following surgery not allowed

    * Vaginal (non-systemic) estrogen allowed
* More than 12 months since prior and no concurrent oral or IV bisphosphonate
* More than 12 months since prior and no concurrent anabolic steroids or growth hormone
* More than 12 months since prior and no concurrent systemic corticosteroids

  * Concurrent short term corticosteroid therapy (to prevent/treat chemotherapy-induced nausea/vomiting) allowed
* More than 6 months since prior and no concurrent Tibolone
* More than 2 weeks since prior and no concurrent drugs known to affect the skeleton (e.g., calcitonin, mithramycin, or gallium nitrate)
* No concurrent chemotherapy or radiotherapy
* No concurrent aromatase inhibitors
* Concurrent enrollment on protocol GOG-0199 allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-11-28 (Actual); Primary Completion 2011-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Alberts, Principal Investigator — Gynecologic Oncology Group
Locations (95):
- United States (95):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Tripler Army Medical Center, Honolulu, Hawaii
  - University of Illinois, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG 0215 accrued 160 patients from November 2005 to April 2010.
Period: Overall Study
Arm/Group | Arm I (Zoledroic Acid) | Arm II (Clinical Observation)
Started | 81 | 79
Completed | 40 | 52
Not Completed | 41 | 27
Not completed — Withdrawal by subject prior to 18 month | 40 | 26
Not completed — Did not have baseline scan | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible and Evaluable subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Zoledroic Acid) | Arm II (Clinical Observation) | Total
Number analyzed (Participants) | 80 | 78 | 158
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 3 | 1 | 4
  30-39 years | 9 | 23 | 32
  40-49 years | 57 | 47 | 104
  50-59 years | 11 | 7 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 78 | 158
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density of the Lumbar Spine as Measured by Dual-energy X-ray Absorptiometry (DEXA) Scan at 9 Months
Description: To compare the effect of zoledronic acid administered every 6 months on bone loss associated with surgery (at a minimum, any surgical procedure that results in removal of both ovaries), as compared with observation alone. This is to be evaluated by measuring the change from baseline to 9 months in bone mineral density (BMD) of the lumbar spine, specifically L1-L4 dual energy X-ray absorptiometry (DEXA).
Time Frame: 9 Months
Population: Eligible and Treated Patients
Measure: Mean (Full Range); unit: g/cm2
Arm/Group | Arm I (Zoledroic Acid) | Arm II (Clinical Observation)
Number analyzed (Participants) | 51 | 68
g/cm2 | -0.025 [-0.240 to 0.077] | -0.086 [-0.308 to 0.067]

2. Primary Outcome: Bone Mineral Density of the Lumbar Spine as Measured by Dual-energy X-ray Absorptiometry (DEXA) Scan at 18 Months
Description: To compare the effect of zoledronic acid administered every 6 months on bone loss associated with surgery (at a minimum, any surgical procedure that results in removal of both ovaries), as compared with observation alone. This is to be evaluated by measuring the change from baseline to 18 months in bone mineral density (BMD) of the lumbar spine, specifically L1-L4 dual energy X-ray absorptiometry (DEXA).
Time Frame: 18 months
Population: Eligible and Treated Patients
Measure: Mean (Full Range); unit: g/cm2
Arm/Group | Arm I (Zoledroic Acid) | Arm II (Clinical Observation)
Number analyzed (Participants) | 40 | 52
g/cm2 | -0.001 [-0.199 to 0.093] | -0.094 [-0.349 to 0.280]

3. Primary Outcome: Bone Mineral Density of the Total Hip as Measured by DEXA Scan on Right Hip
Description: To compare the effect of zoledronic acid on the change in BMD of the right hip following treatment, evaluated by measuring the change from baseline to 18 months
Time Frame: 18 months
Population: Eligible and Treated patients
Measure: Mean (Full Range); unit: g/cm2
Arm/Group | Arm I (Zoledroic Acid) | Arm II (Clinical Observation)
Number analyzed (Participants) | 35 | 51
g/cm2 | 0.101 [-0.400 to 1.500] | -0.052 [-0.212 to 0.307]

4. Primary Outcome: Bone Mineral Density of the Total Hip as Measured by DEXA Scan on Left Hip
Description: To compare the effect of zoledronic acid on the change in BMD of the left hip following treatment, evaluated by measuring the change from baseline to 18 months
Time Frame: 18 months
Population: Eligible and Treated patients
Measure: Mean (Full Range); unit: g/cm2
Arm/Group | Arm I (Zoledroic Acid) | Arm II (Clinical Observation)
Number analyzed (Participants) | 40 | 54
g/cm2 | -0.003 [-0.142 to 0.067] | -0.058 [-0.185 to 0.009]

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Arm I (Zoledroic Acid) | Arm II (Clinical Observation)
Serious Adverse Events (participants affected / at risk) | 1/80 | 0/78
Other Adverse Events (participants affected / at risk) | 45/80 | 19/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Zoledroic Acid) (N=80) | Arm II (Clinical Observation) (N=78)
Gastritis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Zoledroic Acid) (N=80) | Arm II (Clinical Observation) (N=78)
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 12 | 0
Rigors/Chills (General disorders) | 14 | 1
Fatigue (General disorders) | 22 | 4
Insomnia (General disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 1
Hot Flashes (Endocrine disorders) | 3 | 6
Hypothyroidism (Endocrine disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Taste Alteration (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 0
Anorexia (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 15 | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 0 | 1
Inf Unknown Anc: Sinus (Infections and infestations) | 0 | 1
Edema: Limb (Blood and lymphatic system disorders) | 1 | 1
Creatinine (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mental Status (Nervous system disorders) | 1 | 0
Mood Alteration - Depression (Nervous system disorders) | 0 | 3
Mood Alteration - Anxiety (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1
Neuropathy-Sensory (Nervous system disorders) | 1 | 0
Pain - Other (General disorders) | 1 | 1
Pain: Pelvis (General disorders) | 0 | 1
Pain: Vagina (General disorders) | 1 | 1
Pain: Chest /Thorax Nos (General disorders) | 1 | 1
Pain: Head/Headache (General disorders) | 6 | 0
Pain: Neck (General disorders) | 2 | 0
Pain: Extremity-Limb (General disorders) | 0 | 1
Pain: Back (General disorders) | 2 | 1
Pain: Joint (General disorders) | 20 | 4
Pain: Bone (General disorders) | 13 | 1
Pain: Abdominal Pain Nos (General disorders) | 2 | 2
Pain: External Ear (General disorders) | 1 | 0
Pain: Muscle (General disorders) | 19 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Incontinence, Urinary (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 2 | 3
Flu-Like Syndrome (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less